CLINICAL TRIAL: NCT02278614
Title: Efficacy and Safety Assessment of Fixed Combination Unpreserved Latanoprost Eye Drops and Timolol 0.5% (T2347) Versus Xalacom® in Ocular Hypertensive or Glaucomatous Patients.
Brief Title: Efficacy and Safety Assessment of T2347 Versus Xalacom® in Ocular Hypertensive or Glaucomatous Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2347-PIII-12/13
Record Dates: First submitted 2014-10-15; First posted 2014-10-30 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost; Timolol; Xalacom

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2347 (Experimental): T2347: fixed combination Latanoprost 0.005% + Timolol 0.5% unpreserved eye drops
  Interventions: Drug: T2347
- Xalacom (Active Comparator): Xalacom®: Latanoprost 0.005% + Timolol 0.5% preserved eye drops
  Interventions: Drug: Xalacom

INTERVENTIONS:
Drug: T2347 — T2347 eye drop solution is presented in SDU. It is supplied in 0.20 ml single use polyethylene containers.
  Other Names: Latanoprost 0.005% + Timolol 0.5% unpreserved eye drops
  Arms: T2347
Drug: Xalacom — Xalacom® 0.01% eye drop solution is supplied in 2.5 ml multidose container.
  Other Names: Latanoprost 0.005% + Timolol 0.5% preserved eye drops
  Arms: Xalacom

SUMMARY:
The objective of the study is to assess the efficacy and safety of T2347 (Latanoprost 0.005% + Timolol 0.5% unpreserved eye drops) versus Xalacom® in ocular hypertensive or glaucomatous patients initially treated, stabilised by Xalacom® or generics (fixed combination Latanoprost 0.005% + Timolol 0.5% preserved eye drops).

DETAILED DESCRIPTION:
Phase III, international, multicentre, randomised, investigator masked, 3 month duration, 2 parallel groups, 2 X 97 evaluable patients

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent,
* Male or female aged > 18 years old,
* Both eyes with open angle glaucoma or ocular hypertension already treated and controlled by Xalacom® or generics (fixed combination Latanoprost 0.005% + Timolol 0.5% preserved eye drops) since at least 2 months.
* IOP ≤ 18 mmHg in both eyes
* History of IOP insufficiently controlled with first-line monotherapy based on the investigator judgement (e.g. non reaching the target IOP)
* History of an add-on IOP reduction with Xalacom® or generics (fixed combination Latanoprost 0.005% + Timolol 0.5% preserved eye drops) in comparison with first-line treatment
* Corneal thickness ≥ 500 μm and ≤ 600 μm in both eyes.

Exclusion Criteria:

* Ophthalmic exclusion criteria (in either eye)
* Fundoscopy, VF not performed or not available within the 6 months before inclusion visit.
* Significant worsening according to the two last VF (minimum 6 months between these 2 VF)
* Advanced stage of glaucoma:
* Best far corrected visual acuity ≤ 1/10.
* History of trauma, infection, clinically significant inflammation within the 3 months before inclusion visit.
* Ongoing or known history of ocular seasonal and perennial allergy (SAC, PAC) and/or uveitis and/or viral infection.
* Presence of at least one severe objective sign among the following:

  * Hyperaemia (Grade 5)
  * Superficial punctate keratitis (Grade 3)
  * Blepharitis (Grade 3)
* Severe dry eye (defined by severe epithelial erosions of the cornea and/or use of dry eye medication with a frequency exceeding 8 instillations / day).
* Corneal ulceration.
* Palpebral abnormalities not related to medical treatment study and incompatible with a good evaluation.
* History of corneal refractive surgery.
* Any abnormality preventing accurate assessment e.g. reliable tonometry measurement, visual field examination.

Systemic/non ophthalmic exclusion criteria

* Non-controlled diabetic patient.
* Reactive airway disease including bronchial asthma or a history of bronchial asthma, severe chronic obstructive pulmonary disease.
* Sinus bradycardia, sick sinus syndrome, sino-atrial block, second or third degree atrioventricular block not controlled with pace-maker, overt cardiac failure, cardiogenic shock.
* Heart rate <50 bpm, systolic arterial blood pressure≤ 90 mm Hg
* Known or suspected hypersensitivity to one of the components of the study product.
* Any medical or surgical history, disorder or disease such as acute or chronic severe organic disease: hepatic, endocrine, neoplastic, haematological; immunosuppressive, infectious diseases, severe psychiatric illness, relevant cardiovascular abnormalities, etc… and/or any complicating factor or structural abnormality, judged by the investigator to be incompatible with the study.

Specific exclusion criteria for women

* Pregnancy, lactation.
* Childbearing potential woman who is not using a reliable method of contraception

Exclusion criteria related to general conditions

* Inability of patient to understand the study procedures and thus inability to give informed consent.
* Non-compliant patient
* Participation in another clinical study with investigational drug within the last 3 months.
* Already included once in this study.
* Patients being institutionalised because of legal or regulatory order, inmates of psychiatric wards, prison or state institutions, and employees of the study sites or of the Sponsor's company.
* Ward of court.
* Patient not covered by government health care scheme in the country (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, Professor, Principal Investigator — Head of the Glaucoma Clinic
Locations (1):
- Laboratoires Thea, Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2347 | Xalacom
Started | 127 | 115
Completed | 122 | 110
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Adverse Event | 1 | 0
Not completed — left eye was not eligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T2347 | Xalacom | Total
Number analyzed (Participants) | 127 | 115 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 43 | 96
  >=65 years | 74 | 72 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10.8) | 67.2 (10.6) | 66.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 69 | 149
  Male | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of T2347 Compared With Xalacom® on Change in Mean IOP at 9.00 am (± 1 Hour) Between the Baseline (Day 0) and Day 84 in the Worse Eye
Description: the non-inferiority of T2347 unpreserved eye drops compared with Xalacom® on change in mean IOP at 9.00 am (± 1 hour) between the baseline (Day 0) and Day 84 in the worse eye.
  Two relevant time points are considered for this primary criteria: D0 and Day 84.
Time Frame: Day 84
Population: The primary efficacy analysis (mean change in IOP from baseline to Day 84) was performed on the mITT set (236 patients).
  mITT set: All ITT patients with at least one baseline and one post-randomisation efficacy assessment following study treatment.
  242 patients described in the participant flow correpsond to the ITT & Safety set.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | T2347 | Xalacom
Number analyzed (Participants) | 124 | 112
mm Hg | -0.51 (0.18) | -0.52 (0.19)
Statistical Analysis 1: Comparison: T2347 vs Xalacom; Test type: Other — The change from baseline in mean IOP on Day 84 for the contralateral eye,; Mixed Models Analysis; Adjusted mean difference = -0.07, 95% CI 2-sided [-0.57 to 0.43], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: T2347 vs Xalacom; Test type: Other — The change from baseline in mean IOP on D42 for the worse eye; Mixed Models Analysis; Adjusted mean difference = -0.19, 95% CI 2-sided [-0.69 to 0.31], Standard Error of Mean 0.25

ADVERSE EVENTS:
Arm/Group | T2347 | Xalacom
Serious Adverse Events (participants affected / at risk) | 0/127 | 1/115
Other Adverse Events (participants affected / at risk) | 0/127 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2347 (N=127) | Xalacom (N=115)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.